CLINICAL TRIAL: NCT02007070
Title: An Open-label, Non-randomized, Multi-center Phase Ib Study of MK-3475 in Subjects With PD-L1 Positive Advanced Non-small Cell Lung Cancer
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Advanced Non-small Cell Lung Cancer (MK-3475-025/KEYNOTE-025)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-025; 142500 (Registry Identifier: JAPIC-CTI); MK-3475-025 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab 10 mg/kg (Experimental): Participants receive pembrolizumab 10 mg/kg intravenously over 30 minutes on Day 1 of each 21-day cycle for up to 2 years.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous infusion
  Other Names: MK-3475

SUMMARY:
This study is being done to evaluate the safety and efficacy of pembrolizumab (MK-3475) in participants with advanced non-small cell lung cancer (NSCLC) tumors that are positive for programmed cell death ligand 1 (PD-L1): the hypothesis is that treatment with pembrolizumab will result in a clinically meaningful Overall Response Rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC) that is PD-L1 positive per central laboratory review
* At least one measurable lesion
* Radiographic progression of NSCLC after treatment with a platinum-containing doublet for Stage IIIB/IV or recurrent disease
* Eastern Cooperative Oncology Group (ECOG) Performance Scale 0 or 1
* Adequate organ function

Exclusion Criteria:

* Systemic cytotoxic chemotherapy, biological therapy, or major surgery within 3 weeks of the first dose of trial treatment
* Systemic steroid therapy within 3 days prior to the first dose of trial treatment or any other form of immunosuppressive medication
* Expected to require any other form of systemic or localized antineoplastic therapy while on trial
* History of prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or in situ cancer
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease or documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody
* Concurrent or past history of interstitial lung disease
* Pregnant or breast-feeding, or expecting to conceive or father children within the projected duration of the study, starting with screening visit through 120 days after the last dose of pembrolizumab

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Nishio M, Takahashi T, Yoshioka H, Nakagawa K, Fukuhara T, Yamada K, Ichiki M, Tanaka H, Seto T, Sakai H, Kasahara K, Satouchi M, Han SR, Noguchi K, Shimamoto T, Kato T. KEYNOTE-025: Phase 1b study of pembrolizumab in Japanese patients with previously treated programmed death ligand 1-positive advanced non-small-cell lung cancer. Cancer Sci. 2019 Mar;110(3):1012-1020. doi: 10.1111/cas.13932. Epub 2019 Feb 16. PMID 30618179
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with non-small cell lung cancer (NSCLC) who were assessed as being programmed cell death ligand 1 (PD-L1) positive were recruited for this study.
Pre-assignment Details: Thirty-eight (38) participants were enrolled in this study. The data cut-off date for this results disclosure was 30 July 2017.
Groups:
- Pembrolizumab 10 mg/kg: Participants received pembrolizumab 10 mg/kg intravenously over 30 minutes on Day 1 of each 21-day cycle for up to 2 years.
Period: Overall Study
Arm/Group | Pembrolizumab 10 mg/kg
Started | 38
Completed | 5 (Completed 2 years of treatment.)
Not Completed | 33
Not completed — Adverse Event | 4
Not completed — Clinical Progression | 4
Not completed — Death | 1
Not completed — Protocol Violation | 2
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 21

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 26
Programmed Cell Death Ligand 1 (PD-L1) Expression Status [Count of Participants; unit: Participants] — PD-L1 expression was evaluated by immunohistochemistry (IHC) assay with a newly obtained tumor tissue with biopsy. If PD-L1 expression was observed in >1% to ≤50% of tumor cells, regardless of the PD-L1 staining intensity, the participant was defined as weakly positive PD-L1. If PD-L1 expression was observed in >50% of tumor cells, the participant was defined as strongly positive PD-L1.
  Participants
    Strongly Positive PD-L1 | 12
    Weakly Positive PD-L1 | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Strongly PD-L1 Positive Participants
Description: On-study imaging was to be performed every 9 weeks after the first dose of study drug, or more frequently if clinically indicated. ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters). The percentage of strongly PD-L1 positive participants who experienced a CR or PR is presented.
Time Frame: Up to 2 years
Population: The Full Analysis Set (FAS) population consisted of all participants who were classified as strongly PD-L1 positive, received at least one dose of study drug and had Baseline data for the analyses that required Baseline data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 11
Percentage of Participants | 27.3 [6.0 to 61.0]

2. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of the study drug, was also an AE. After discontinuation of study drug, each participant was monitored for a minimum of 30 days for AE monitoring (serious AEs were monitored for up to 90 days after last dose of study drug). The number of participants who experienced an AE is presented.
Time Frame: Up to 27 months (Up to 90 days after last dose of study drug)
Population: The All Treated Set (ATS) population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 38
Participants | 38

3. Primary Outcome: Number of Participants Discontinuing Study Drug Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of the study drug, was also an AE. The number of participants who discontinued study drug due to an AE is presented.
Time Frame: Up to 2 years
Population: The ATS population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 38
Participants | 4

4. Secondary Outcome: Progression Free Survival (PFS) by RECIST 1.1 in Strongly PD-L1 Positive Participants
Description: PFS was defined as the time from the first day of study treatment to the first documented disease progression per RECIST 1.1 based on blinded independent central radiologists' review or death due to any cause, whichever occurred first. Using RECIST 1.1, progressive disease was defined as either a 20% relative increase in the sum of diameters of target lesions, taking as reference the smallest sum on study OR an absolute increase of >5 mm in the sum of lesions, OR the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and is reported in months. The median PFS for all strongly PD-L1 positive participants is presented.
Time Frame: Up to 2 years
Population: The ATS population for this outcome measure consisted of all strongly PD-L1 positive participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 12
Months | 4.1 [1.6 to 19.1]

5. Secondary Outcome: Duration of Response (DOR) by RECIST 1.1 in Strongly PD-L1 Positive Participants
Description: DOR was measured from the time measurement criteria were first met for CR/PR (whichever was first recorded) until the first date that recurrent or progressive disease was objectively documented (taking as reference for progressive disease the smallest measurements recorded on study). DOR was censored at the last tumor assessment date if a responder did not have PD or death. Non-responders were not included in the analysis. The lower and upper limits were estimated at the time of data cutoff. DOR was analyzed using the Kaplan-Meier method and is reported in days. The median DOR for all strongly PD-L1 positive participants with a confirmed response is presented.
Time Frame: Up to 2 years
Population: The ATS population for this outcome measure consisted of all strongly PD-L1 positive participants who received at least one dose of study drug and experienced a confirmed response.
Measure: Median (Full Range); unit: Days
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 3
Days | NA [454.0 to NA] — Median DOR not reached. For upper limit, no progressive disease by the time of last disease assessment.

6. Secondary Outcome: Overall Survival (OS) in Strongly PD-L1 Positive Participants
Description: OS was defined as the time from the first day of study treatment to death due to any cause. OS is reported for all strongly PD-L1 positive participants in months
Time Frame: Up to 2 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 12
Months | 17.9 [5.9 to NA] — Upper limit not reached.

7. Secondary Outcome: ORR Per Immune-Related Response Criteria (irRC) in Strongly PD-L1 Positive Participants
Description: ORR per irRC was defined as the percentage of participants in the analysis population who had a Complete Response (irCR: Complete disappearance of all tumor lesions [whether measureable or not, and no new lesions; irCR must be confirmed by repeated, consecutive assessments made no less than 4 weeks from the date first documented]) or Partial Response (irPR: Decrease in sum of the products of the two largest perpendicular diameters [SPD] of 50% or greater by a consecutive assessment at least 4 weeks after first documentation). The percentage of strongly PD-L1 positive participants who experienced an irCR or irPR is presented.
Time Frame: Up to 2 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 12
Percentage of Participants | 25.0 [5.5 to 57.2]

8. Secondary Outcome: PFS Per irRC in Strongly PD-L1 Positive Participants
Description: PFS was defined as the time from the first day of study treatment to the first documented disease progression per irRC or death due to any cause, whichever occurred first. Using irRC, progressive disease was defined as at least a 25% increase in SPD relative to minimum recorded tumor burden. Confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented was required. Median PFS was analyzed using the Kaplan-Meier method and is presented in months for all strongly PD-L1 positive participants.
Time Frame: Up to 2 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 12
Months | 5.2 [2.8 to 12.5]

9. Secondary Outcome: DOR Per irRC in Strongly PD-L1 Positive Participants
Description: DOR was measured from the time measurement criteria were first met for irCR/irPR (whichever was first recorded) until the first date that recurrent or progressive disease (PD) was objectively documented (taking as reference for progressive disease the smallest measurements recorded on study). PD was defined as at least a 25% increase in SPD relative to minimum recorded tumor burden. Confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented was required. DOR was censored at the last tumor assessment date if a responder did not have PD or death. Non-responders were not included in the analysis. DOR was analyzed using the Kaplan-Meier method, is reported in days and is presented for all strongly PD-L1 positive participants who experienced an irCR or irPR.
Time Frame: Up to 2 years
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 3
Days | 503.0 [127.0 to NA] — For upper limit, no progressive disease by the time of last disease assessment.

10. Secondary Outcome: ORR Per RECIST 1.1 in PD-L1 Positive Participants
Description: On-study imaging was to be performed every 9 weeks after the first dose of study drug, or more frequently if clinically indicated. ORR was defined as the percentage of participants in the analysis population who had a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters). The percentage of PD-L1 positive participants who experienced a CR or PR is presented.
Time Frame: Up to 2 years
Population: The FAS population for this outcome measure consisted of all participants who were classified as PD-L1 positive, received at least one dose of study drug and had Baseline data for the analyses that required Baseline data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 37
Percentage of Participants | 21.6 [9.8 to 38.2]

11. Secondary Outcome: PFS by RECIST 1.1 in PD-L1 Positive Participants
Description: PFS was defined as the time from the first day of study treatment to the first documented disease progression per RECIST 1.1 based on blinded independent central radiologists' review or death due to any cause, whichever occurred first. Using RECIST 1.1, progressive disease was defined as either a 20% relative increase in the sum of diameters of target lesions, taking as reference the smallest sum on study OR an absolute increase of >5 mm in the sum of lesions, OR the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and is reported in months. The median PFS for all PD-L1 positive participants is presented.
Time Frame: Up to 2 years
Population: The ATS population for this outcome measure consisted of all PD-L1 positive participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 38
Months | 3.9 [2.0 to 6.2]

12. Secondary Outcome: DOR by RECIST 1.1 in PD-L1 Positive Participants
Description: DOR was measured from the time measurement criteria were first met for CR/PR (whichever was first recorded) until the first date that recurrent or progressive disease was objectively documented (taking as reference for progressive disease the smallest measurements recorded on study). DOR was censored at the last tumor assessment date if a responder did not have PD or death. Non-responders were not included in the analysis. The lower and upper limits were estimated at the time of data cutoff. DOR was analyzed using the Kaplan-Meier method and is reported in days. The median DOR for all PD-L1 positive participants with a confirmed response is presented.
Time Frame: Up to 2 years
Population: The ATS population for this outcome measure consisted of all PD-L1 positive participants who received at least one dose of study drug and experienced a confirmed response.
Measure: Median (Full Range); unit: Days
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 8
Days | 694.0 [120.0 to NA] — For upper limit, no progressive disease by the time of last disease assessment.

13. Secondary Outcome: OS in PD-L1 Positive Participants
Description: OS was defined as the time from the first day of study treatment to death due to any cause. OS is reported for all PD-L1 positive participants in months.
Time Frame: Up to 2 years
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 38
Months | 19.2 [8.0 to 26.7]

14. Secondary Outcome: ORR Per irRC in PD-L1 Positive Participants
Description: ORR per irRC was defined as the percentage of participants in the analysis population who had a irCR (Complete disappearance of all tumor lesions [whether measureable or not, and no new lesions; irCR must be confirmed by repeated, consecutive assessments made no less than 4 weeks from the date first documented]) or irPR (Decrease in sum of the products of the two largest perpendicular diameters [SPD] of 50% or greater by a consecutive assessment at least 4 weeks after first documentation). The percentage of PD-L1 positive participants who experienced an irCR or irPR is presented.
Time Frame: Up to 2 years
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 38
Percentage of Participants | 21.1 [9.6 to 37.3]

15. Secondary Outcome: PFS Per irRC in PD-L1 Positive Participants
Description: PFS was defined as the time from the first day of study treatment to the first documented disease progression per irRC or death due to any cause, whichever occurred first. Using irRC, progressive disease was defined as at least a 25% increase in SPD relative to minimum recorded tumor burden. Confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented was required. Median PFS was analyzed using the Kaplan-Meier method and is presented in months for all PD-L1 positive participants.
Time Frame: Up to 2 years
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 38
Months | 4.2 [3.4 to 7.6]

16. Secondary Outcome: DOR Per irRC in PD-L1 Positive Participants
Description: DOR was measured from the time measurement criteria were first met for irCR/irPR (whichever was first recorded) until the first date that recurrent or progressive disease (PD) was objectively documented (taking as reference for progressive disease the smallest measurements recorded on study). PD was defined as at least a 25% increase in SPD relative to minimum recorded tumor burden. Confirmation by a repeat, consecutive assessment no less than 4 weeks from the data first documented was required. DOR was censored at the last tumor assessment date if a responder did not have PD or death. Non-responders were not included in the analysis. DOR was analyzed using the Kaplan-Meier method, is reported in days and is presented for all PD-L1 positive participants who experienced an irCR or irPR.
Time Frame: Up to 2 years
Population: as for outcome 12
Measure: Median (Full Range); unit: Days
Arm/Group | Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 8
Days | 757.0 [120.0 to NA] — For upper limit, no progressive disease by the time of last disease assessment.

ADVERSE EVENTS:
Time Frame: Up to 27 months (Up to 90 days after last dose of study drug)
Description: The ATS population consisted of all participants who received at least one dose of study drug.
Arm/Group | Pembrolizumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/38
Serious Adverse Events (participants affected / at risk) | 14/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 10 mg/kg (N=38)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 10 mg/kg (N=38)
Anaemia (Blood and lymphatic system disorders) | 2 (5)
Hypothyroidism (Endocrine disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (9)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (7)
Periodontal disease (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 5 (6)
Injection site reaction (General disorders) | 2 (2)
Malaise (General disorders) | 9 (12)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 11 (14)
Bronchitis (Infections and infestations) | 3 (4)
Conjunctivitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 8 (8)
Blood alkaline phosphatase increased (Investigations) | 7 (7)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 5 (5)
Lymphocyte count decreased (Investigations) | 5 (6)
Platelet count decreased (Investigations) | 2 (2)
Weight decreased (Investigations) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (6)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 6 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (12)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.